CLINICAL TRIAL: NCT00004428
Title: Phase I Randomized Study of CPX for the Treatment of Adult Patients With Mild Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: SciClone Pharmaceuticals (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13364; SCICLONE-FDA-OP-97-1
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-01

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases

INTERVENTIONS:
Drug: CPX

SUMMARY:
OBJECTIVES: I. Evaluate the safety of ascending doses of CPX administered to adult patients with mild cystic fibrosis.

II. Evaluate the pharmacokinetics of ascending doses of CPX in this patient population.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, dose escalation study.

There are 7 experimental cohorts, each treated with a different oral dose of CPX or placebo. Within each cohort, 4 patients receive a single dose of CPX and 1 patient receives placebo. Each patient is monitored 24 hours postdose. Escalation to the next dose level for each subsequent cohort begins only after the safety data obtained from the previous cohort is reviewed and found not to limit dose escalation.

All patients return for a follow up evaluation 1 week after dosing.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Mild cystic fibrosis
* Not pregnant or nursing Negative pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 1997-09; Study Completion 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Martins, Study Chair — SciClone Pharmaceuticals

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662